CLINICAL TRIAL: NCT00999375
Title: Cultivating Healthy Environments in Families With Type 1 Diabetes (CHEF)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 999909234; 09-CH-N234
Record Dates: First submitted 2009-10-20; First posted 2009-10-21 (Estimated); Last update posted 2019-11-29 (Actual); Status verified 2019-10-30

CONDITIONS: Type I Diabetes
Keywords: Type 1 Diabetes; Diet; Behavioral Intervention; Children; Adolescents
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Educational Status; Behavior Therapy

ARMS (2):
- Group A (Experimental)
  Interventions: Behavioral: Education; Behavioral: Problem Solving; Behavioral: Social Learning; Behavioral: Behavior Modification
- Group B (Active Comparator)
  Interventions: Behavioral: Education

INTERVENTIONS:
Behavioral: Education
Behavioral: Problem Solving
  Arms: Group A
Behavioral: Social Learning
  Arms: Group A
Behavioral: Behavior Modification
  Arms: Group A

SUMMARY:
Background:

* Type 1 diabetes (T1D) is a common chronic disease in children, occurring in approximately 1 of every 400 to 600 children. Children with T1D are unable to produce insulin, a hormone that allows the body to use glucose from food. Children with T1D manage their diabetes by taking insulin, monitoring their blood glucose levels, and watching their diet, including carbohydrates.
* Carbohydrates come from many different kinds of food, and recent research has shown that different foods have a different effect on the level of glucose in the blood. In general, whole, unprocessed foods (e.g., fruits, vegetables, whole grains, legumes) have a lower glycemic index (GI), which means that they cause smaller, more sustained blood sugar levels. Additionally, these foods are rich in nutrients. Nutrient-poor carbohydrates come from foods made with refined grains and sugars, such as breads, crackers, and breakfast cereals; they general cause a more rapid increases in blood sugar (i.e., a high GI). Lower GI diets may help people with T1D manage their blood glucose levels more easily.

Objectives:

* To determine the utility of a whole foods, low GI diet in the management of T1D.
* To determine the utility of a behavioral intervention to promote healthful family dietary behaviors, including eating more fruits, vegetables, whole grains, and legumes, and fewer refined carbohydrates.
* To determine how the dietary intervention affects quality of life, satisfaction with the diet, and risk for problem eating behaviors.

Eligibility:

- Children 8 to 16 years of age who have been diagnosed with T1D for more than 12 months, and who use insulin injections to maintain normal blood glucose levels.

Design:

* Families will be divided into two groups: an intervention group that will participate in intensive dietary intervention and continuous glucose monitoring (CGM) and a control group that will not have the dietary intervention but will have CGM and scheduled contacts with study staff.
* Intervention group families will have 11 family-based and 2 group-based sessions consisting of behavioral techniques and educational content about eating nutrient-dense, low GI foods. CGM results will give families feedback about how their diet affects blood glucose levels. At least one parent and the child with T1D will participate in the intervention.
* Intervention topics will consist of goal setting, behavior self-monitoring, educational information, and problem solving, among others. Parents and children will record the foods they eat.
* Control group families will participate in 11 family-based sessions consisting of CGM feedback.
* Assessments will be conducted at 6, 12, and 18 months, and medical record information, including blood and urine testing, will be obtained at each routine clinic visit.

DETAILED DESCRIPTION:
This protocol describes a randomized controlled trial to promote consumption of carbohydrates from nutrient-dense whole foods among children and adolescents with type 1 diabetes and to determine the efficacy of such dietary changes in improving glycemic control and other diabetes-related health outcomes.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Child age 8.0-16.9 years
  2. T1D: classical presentation and/or antibody positivity
  3. Diabetes duration greater than or equal to 12 months
  4. Daily insulin dose greater than or equal to 0.5 units/kilogram
  5. Hemoglobin A1c greater than or equal to 7.0% and less than or equal to 9.5%
  6. Insulin regimen

     * a. Greater than or equal to 3 injections daily, OR
     * b. Continuous subcutaneous insulin infusion (insulin pump) (CSII)
  7. Blood glucose monitoring frequency: Greater than or equal to 3 checks daily
  8. Stable living situation (guardian and address) for greater than or equal to 6 months
  9. Joslin Clinic attendance

     * a. At least one Joslin Clinic visit in last year, AND
     * b. Anticipated care at Joslin Clinic for duration of study

EXCLUSION CRITERIA:

1. Daily use of premixed insulin
2. Transition to CSII (insulin pump) therapy in last 3 months
3. Continuous glucose monitoring use in last 3 months
4. Participation in a different intervention study in the last 6 months
5. Presence of co-morbid conditions (any of the following):

   * a. Celiac disease, inflammatory bowel disease, or other significant gastrointestinal condition
   * b. Systemic glucocorticoid use (cumulative 1 month during last year)
   * c. Significant multiple food allergies
   * d. Significant mental illness defined by either:

     * 1. Major psychiatric disorder (e.g., eating disorder, major psychoses), OR
     * 2. Inpatient psychiatric admission during last 6 months
6. Significant medical or psychiatric illness in caregiver that would prevent active participation in the study
7. Intent to enroll in another intervention study during the course of this study

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 293 (Actual)
Dates: Start 2009-09-18; Primary Completion 2013-11-27 (Actual); Study Completion 2013-11-27 (Actual)

PRIMARY OUTCOMES:
Change in glycemic control, change in dietary intake | 18 months

SECONDARY OUTCOMES:
Change in social cognitive mediators of behavior; change in psychosocial status; change in body composition, lipids, oxidative stress, and inflammation

CONTACTS AND LOCATIONS:
Overall Officials: Tonja R. Nansel, Ph.D., Principal Investigator — Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD)
Locations (1):
- Joslin Diabetes Center, Boston, Massachusetts, United States

REFERENCES:
- [Background] American Diabetes Association. Nutrition Recommendations and Interventions for Diabetes: a position statement of the American Diabetes Association. Diabetes Care. 2007 Jan;30 Suppl 1:S48-65. doi: 10.2337/dc07-S048. No abstract available. PMID 17192379
- [Background] Anderson BJ, Auslander WF, Jung KC, Miller JP, Santiago JV. Assessing family sharing of diabetes responsibilities. J Pediatr Psychol. 1990 Aug;15(4):477-92. doi: 10.1093/jpepsy/15.4.477. PMID 2258796
- [Background] Anderson EJ, Richardson M, Castle G, Cercone S, Delahanty L, Lyon R, Mueller D, Snetselaar L. Nutrition interventions for intensive therapy in the Diabetes Control and Complications Trial. The DCCT Research Group. J Am Diet Assoc. 1993 Jul;93(7):768-72. doi: 10.1016/0002-8223(93)91750-k. PMID 8320402
- [Derived] Ortiz La Banca Barber R, Volkening LK, Mehta SN, Dassau E, Laffel LM. Effects of Macronutrient Intake and Number of Meals on Glycemic Outcomes Over 1 Year in Youth with Type 1 Diabetes. Diabetes Technol Ther. 2024 Jun;26(6):420-425. doi: 10.1089/dia.2023.0464. Epub 2024 Feb 13. PMID 38277162
- [Derived] Sanjeevi N, Lipsky L, Liu A, Nansel T. Differential reporting of fruit and vegetable intake among youth in a randomized controlled trial of a behavioral nutrition intervention. Int J Behav Nutr Phys Act. 2019 Feb 1;16(1):15. doi: 10.1186/s12966-019-0774-9. PMID 30709403
- [Derived] Lipsky LM, Haynie DL, Liu A, Nansel TR. Resemblance of Diet Quality in Families of Youth with Type 1 Diabetes Participating in a Randomized Controlled Behavioral Nutrition Intervention Trial in Boston, MA (2010-2013): A Secondary Data Analysis. J Acad Nutr Diet. 2019 Jan;119(1):98-105. doi: 10.1016/j.jand.2018.07.025. Epub 2018 Oct 31. PMID 30389377
- [Derived] Quick V, Lipsky LM, Nansel TR. Psychometric properties and factor structure of the adapted Self-Regulation Questionnaire assessing autonomous and controlled motivation for healthful eating among youth with type 1 diabetes and their parents. Child Care Health Dev. 2018 Jul;44(4):651-658. doi: 10.1111/cch.12574. Epub 2018 May 16. PMID 29770461
- [Derived] Nansel TR, Lipsky LM, Haynie DL, Eisenberg MH, Dempster K, Liu A. Picky Eaters Improved Diet Quality in a Randomized Behavioral Intervention Trial in Youth with Type 1 Diabetes. J Acad Nutr Diet. 2018 Feb;118(2):308-316. doi: 10.1016/j.jand.2017.10.012. PMID 29389510
- [Derived] Eisenberg Colman MH, Quick VM, Lipsky LM, Dempster KW, Liu A, Laffel LMB, Mehta SN, Nansel TR. Disordered Eating Behaviors Are Not Increased by an Intervention to Improve Diet Quality but Are Associated With Poorer Glycemic Control Among Youth With Type 1 Diabetes. Diabetes Care. 2018 Apr;41(4):869-875. doi: 10.2337/dc17-0090. Epub 2018 Jan 25. PMID 29371234
- [Derived] Nansel TR, Lipsky LM, Eisenberg MH, Liu A, Mehta SN, Laffel LM. Can Families Eat Better Without Spending More? Improving Diet Quality Does Not Increase Diet Cost in a Randomized Clinical Trial among Youth with Type 1 Diabetes and Their Parents. J Acad Nutr Diet. 2016 Nov;116(11):1751-1759.e1. doi: 10.1016/j.jand.2016.07.005. Epub 2016 Aug 31. PMID 27597745
- [Derived] Nansel TR, Lipsky LM, Liu A. Greater diet quality is associated with more optimal glycemic control in a longitudinal study of youth with type 1 diabetes. Am J Clin Nutr. 2016 Jul;104(1):81-7. doi: 10.3945/ajcn.115.126136. Epub 2016 May 18. PMID 27194309
- [Derived] Widaman AM, Witbracht MG, Forester SM, Laugero KD, Keim NL. Chronic Stress Is Associated with Indicators of Diet Quality in Habitual Breakfast Skippers. J Acad Nutr Diet. 2016 Nov;116(11):1776-1784. doi: 10.1016/j.jand.2016.03.016. Epub 2016 May 6. PMID 27161025
- [Derived] Nansel TR, Laffel LM, Haynie DL, Mehta SN, Lipsky LM, Volkening LK, Butler DA, Higgins LA, Liu A. Improving dietary quality in youth with type 1 diabetes: randomized clinical trial of a family-based behavioral intervention. Int J Behav Nutr Phys Act. 2015 May 8;12:58. doi: 10.1186/s12966-015-0214-4. PMID 25952160